CLINICAL TRIAL: NCT05230095
Title: Social Cognition Dysfunctions in Parkinson's Disease
Acronym: cognition 2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1154; 2022-A00216-37 (Other: ID-RCB)
Record Dates: First submitted 2022-01-28; First posted 2022-02-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; emotional recognition; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's disease patients: 30 parkinsonian patients scheduled for deep brain stimulation implantation surgery will be recruited
  Interventions: Behavioral: social cognition tests; Behavioral: Quality of life self-questionnaire
- Controls: 15 healthy volunteers matched in age and sex will be recruited
  Interventions: Behavioral: social cognition tests

INTERVENTIONS:
Behavioral: social cognition tests — The evaluation of social cognition will be carried out using questionnaires and a point lights computer test. During the computer test, participants have to watch several short sequences of interactions between two silhouettes and give an interpretation of the scene.
  Patients will be evaluated twice: one time before the surgery and a second time 1 year after surgery.
  Healthy volunteers will be evaluated only one time.
Behavioral: Quality of life self-questionnaire — Quality of life will be assessed using a self-administered questionnaire in the patients group only.
  Groups: Parkinson's disease patients

SUMMARY:
Parkinson's disease (PD) is usually responsible of cognitive and behavioral non-motor signs with a major impact on the quality of life. Social cognition is a complex system relying on emotion recognition (neurons mirror system (NMS)), the theory of mind (with its two parts: emotional and cognitive), but also on the social and cultural environment and the personal history. The first step in this model is represented by the NMS, which seems to be altered in PD patients for both positive and negative emotions as shown in our preliminary study. The investigator purpose is to investigate the role of the treatment (levodopa and deep brain stimulation) on the functioning of the NMS

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Man or woman
* Participant not objecting to participation in the study
* Age ≥ 30 and ≤ 70 years old

Specific inclusion criteria for patients:

* Patients with Parkinson's disease with motor fluctuations and dyskinesias receiving deep-brain stimulation
* Patients able to understand the issues of the study

Exclusion Criteria:

For all participants:

* Person deprived of liberty by judicial or administrative decision
* Person subject to a legal protection measure (tutorship, curatorship)
* Person concurrently participating in another research project who may interfere with the results or conclusions of this study

Specific exclusion criteria for healthy volunteers

* Person presenting or having presented a neurological or psychiatric pathology
* Person with a serious medical condition
* Person who has exceeded the annual amount of compensation authorized for participation in research protocols

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients likely to participate in the study and verifying the eligibility criteria will be identified within the Neurology C department as part of their neurological follow-up before and after deep brain stimulation.
  Healthy volunteers will be recruited among the spouses of the patients or via association like France Parkinson.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

PRIMARY OUTCOMES:
Emotional resonance task score | 12 months following the inclusion
  In the emotional resonance task, patients are asked to rate the emotional valence of fifteen 3-second silent videos. These movies show emotionally connoted motor interactions between two persons, each of them being depicted by 20 white dots moving on a black background (Point Light Displays (PLD) technique). Among these 15 videos, 5 has a negative valence (making someone cry, sadness, argument, hitting someone and anger), 5 has a positive valence (joy, dancing, giving a flower, laughing and cuddling) and 5 neutral valences (sit, stand, say hello, raise your arms and saw).
  The Emotional resonance score in parkinsonian patients undergoing treatment (dopaminergic or deep brain stimulation) will be compared to their score without treatment (OFF Dopa or OFF stimulation).

SECONDARY OUTCOMES:
Correlations between the emotional resonance task score and patients' quality of life self-questionnaire score (PDQ39) | 12 months following the inclusion
  PDQ39 (Parkinson's Disease Questionnaire) is a 39-item self-report questionnaire assessing Parkinsons' disease-specific health and well-being over the last month. PDQ39 provide a summary score of the impact of the illness on functioning and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurology C department, P. Wertheimer Hospital, Bron, France